CLINICAL TRIAL: NCT02193802
Title: Role of Capsule Endoscopy in the Evaluation of Mucosal Changes During Treatment of Patients With Active Crohn's Disease
Acronym: CHANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GETAID 2012-3; 2013-A00034-41 (Other: ANSM (french regulatory authority))
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; small bowel (SB); capsule endoscopy; ileocolonoscopy; anti-TNF-alpha antibodies
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopy (Other): CHANCE is a single arm study: all patients will undergo one capsule endoscopy ( PillCam® COLON 2 capsule and PillCam Crohn's) of the whole intestine AND one ileocolonoscopy.
  The patients will be then treated according to the preference of their physician and a second capsule endoscopy AND an ileoconoscopy will be performed 6 at 12 months later.
  Both exams will be evaluated locally by two independent investigators and all the recorded films will be evaluated and compared by four central readers.
  Interventions: Device: PillCam® COLON 2 and PillCam Crohn's capsules

INTERVENTIONS:
Device: PillCam® COLON 2 and PillCam Crohn's capsules — Patient preparation for PillCam® COLON 2 and PillCam Crohn's capsule procedure:
  Patients will drink only clear liquids beginning 12 noon the day prior to the procedure,12 hour fast prior to the procedure and 1 L of PEG on the morning two hours before the capsule ingestion.
  Patients can drink clear liquids 2 hours and eat 4 hours post ingestion. Eight hours post ingestion the data recorder should be removed. Patients will confirm excretion of the capsule or as required by the investigator.

SUMMARY:
The utility of capsule endoscopy in diagnosing small bowel (SB) Crohn's disease has been demonstrated in a number of studies.

Mucosal healing is a good predictor of long term remission. Unfortunately, the assessment of small bowel mucosal healing by conventional colonoscopy is an invasive technique which is not complete since it does not allow exploration of the small bowel beyond the terminal ileum (TI). Thus, direct evidence of the healing of the majority of the small bowel is lacking.

DETAILED DESCRIPTION:
Crohn's disease is a chronic, inflammatory disorder affecting any part of the gastrointestinal tract but the terminal ileum is the most frequent location involved alone or in combination with other locations. While about one half of patients have involvement of the ileum and large bowel, another third have disease limited to the small bowel.

The disease affects populations around the globe and occurs at any age but tends to have a peak incidence between the ages of 15 and 35. Typical presenting symptoms include abdominal pain and diarrhea. The clinical presentation of Crohn's disease fluctuates throughout the course of the disease. Symptoms and signs usually correlate with mucosal inflammation. The pattern of Crohn's disease viewed on endoscopy has been characterized and is associated with a number of mucosal characteristics such as erythema, swelling, nodularity, strictures, aphthoid ulceration and ulcers of variable size and depth.

The utility of capsule endoscopy in diagnosing small bowel (SB) Crohn's disease has been demonstrated in a number of studies. Diagnostic yields of 70% have been reported in suspected SB Crohn's disease. In patients with a known Crohn's disease, the superiority of the capsule to detect mucosal lesions of the SB in comparison to any other radiologic technique has also been clearly demonstrated.

A number of studies indicate that mucosal healing is a good predictor of long term remission. In particular, intense therapeutic regimens including purine analogues and biologic therapies like infliximab have been associated with endoscopic mucosal healing. The recently published SONIC trial evaluated the efficacy of infliximab monotherapy, azathioprine monotherapy and the two drugs combined in moderate to severe Crohn's disease patients. Patients who were treated with infliximab monotherapy and with the combination therapy had significantly longer corticosteroid-free clinical remission than those receiving azathioprine alone. Furthermore, mucosal healing, defined as the absence of mucosal ulcerations at week 26, was greater for the combination therapy than each of the monotherapies alone. Based on the results of these studies, obtaining a mucosal healing becomes in clinical practice a new therapeutic objective especially in patients treated by immunosuppressors or anti-TNF-alpha antibodies. In most of the studies, a complete mucosal healing was assessed by the complete disappearance of ulceration. An endoscopic response could be evaluated by the variation of several endoscopic scores of severity, that are either dedicated to the terminal ileon (TI) more the colon i.e. the Crohn's disease endoscopic severity index (CDEIS) or to the SB i.e. the Lewis score. Concerning the evaluation of the mucosal lesions of the SB by the capsule, a new index of severity is being developed in a study conducted by the different centers of the GETAID i.e. the CE-CDEIS. This score will be available in the first semester of 2013 and would be usable for the present study.

Unfortunately, the assessment of mucosal healing by conventional ileocolonoscopy is not complete since it does not allow exploration of the small bowel beyond TI. Thus, while mucosal changes and symptomatic improvement in subjects with SB Crohn's disease (with or without colonic involvement) can be inferred from studies like ACCENT I, direct evidence of the healing of the majority of the small bowel is lacking. In addition, correlation between evidence of mucosal healing and symptoms, as measured by the Crohn's Disease Activity Index (CDAI), has not been found reliable. This may reflect the limitation of viewing the full extent of small bowel ulcerations on the limited examination which is possible with ileocolonoscopy. This may potentially be overcome with the use of capsule endoscopy of the small bowel.

Until now, no study has evaluated the potential treatment-induced changes of the mucosal lesions located in the SB with a capsule and no comparison between the capsule and the ileocolonoscopy has been conducted in the evaluation of the TI which is the segment analyzable by both techniques. For the patients, demonstrate that the capsule is usable to evaluate the mucosal healing, would be a considerable benefit knowing that the capsule do not necessitate an arduous bowel cleansing and a sedation or a general anesthesia.

The proposed study is designed as a pilot study to evaluate the role of capsule endoscopy in Crohn's disease patients, in monitoring the changes in the terminal ileum and small bowel mucosa during Crohn's disease treatment for induction of remission in active Crohn's disease with ileal involvement. Success in this trial may lead to a larger trial to validate the findings.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged more than 18 years
* Subject with at least ileal lesions of Crohn's disease
* Subject with moderate to severe Crohn's disease at baseline, as defined by CDAI > 150,
* Subject accepting to undergo two capsules endoscopy and Ileocolonoscopy procedures
* Proven patency by Agile capsule or another approach deemed clinically acceptable by the investigator, e.g. CT enterography or MRI enterography, performed within the 6 months prior to enrollment

Exclusion Criteria:

* Known gastrointestinal obstruction or strictures based on the clinical picture or pre procedure testing and profile
* Cardiac pacemakers or other implanted electromedical devices
* Swallowing disorders.
* Subject with known slow gastric emptying
* Contraindications to ileocolonoscopy or general anasthesia
* Subject with any condition, which precludes compliance with study and/or device instructions
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study
* Subject has taken NSAID medications less than one month before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the agreement between capsule and ileocolonoscopy in the change of physician global assessment (PGA) as visualized in the TI in patients under treatment. | week 0 and after 6 at 12 months
  PGA will be evaluated based on capsule or Ileocolonoscopy procedures at week 0 and after 6 at 12 months in two ways as follows:
  Quantitative PGA assessment: the severity of the disease will be graded on an analogue visual scaled from 0 (no lesions identified) to 10 (lesions of maximum severity identified).
  Qualitative PGA assessment: the severity of the disease at weeks 0 and 40 will be classified into one of the following categories:
  * No active disease
  * Mild disease
  * Moderate disease
  * Severe disease
  Physician global assessment of the disease severity variation will be classified into:
  * Definite Improvement
  * Slightly improvement
  * No change
  * Slightly worsening
  * Definite Worsening
  Disease severity variation will be also quantified by the change in quantitative PGA.
  The disease global severity will be later estimated by the two independent local investigators based on the previously capsule small bowel PGA and on the colonoscopy previously colon PGA.

SECONDARY OUTCOMES:
Lewis score | week 0 and after 6 at 12 months
  The local readers will categorize lesions identified in RAPID. The Lewis score will be calculated later using a dedicated feature in the Rapid software, where the outcome is a continuous scale variable.
Segmental ileal and global CDEIS score | week 0 and after 6 at 12 months
  Segmental ileal and global CDEIS score will be evaluated later in continuance way based on ileo-colonoscopy and capsule findings at weeks 0 and after 6 at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Arnaud Bourreille, MD, Principal Investigator — CHU Nantes, Service Hépato-gastro-entérologie 1, place Alexis Ricordeau 44093 Nantes Cedex 1
Locations (11):
- France (10):
  - CHU Amiens, Amiens
  - CHU CAEN, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Huriez, Lille
  - Hôpital Brabois, Nancy
  - Hôpital Hôtel Dieu, Nantes
  - Hôpital Archet 2, Nice
  - Hôpital St Louis, Paris
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Background] Sands B.E. Crohn's Disease. Sleisenger and Fortran's Gastrointestinal and Liver Disease. 8th edition; Volume 2; Saunders Elsevier Publisher; Canada. 2006. pps 2459-2498.
- [Background] Lichtenstein G.R. The Clinician's Guide to Inflammatory Bowel Disease. Slack Publishers, New Jersey 2003. pps 1-7;16-19; 41-57.
- [Background] Kornbluth A, Colombel JF, Leighton JA, Loftus E; ICCE. ICCE consensus for inflammatory bowel disease. Endoscopy. 2005 Oct;37(10):1051-4. doi: 10.1055/s-2005-870315. No abstract available. PMID 16189789
- [Background] Engstrom P.F. Goosenberg E.B. Diagnosis and Management of Bowel Disease. 1st edition. Professional Communications, Inc. Publisher. Oklahoma. 1999. pps. 169-185.
- [Background] Sipponen T, Savilahti E, Kolho KL, Nuutinen H, Turunen U, Farkkila M. Crohn's disease activity assessed by fecal calprotectin and lactoferrin: correlation with Crohn's disease activity index and endoscopic findings. Inflamm Bowel Dis. 2008 Jan;14(1):40-6. doi: 10.1002/ibd.20312. PMID 18022866
- [Background] Sostegni R, Daperno M, Scaglione N, Lavagna A, Rocca R, Pera A. Review article: Crohn's disease: monitoring disease activity. Aliment Pharmacol Ther. 2003 Jun;17 Suppl 2:11-7. doi: 10.1046/j.1365-2036.17.s2.17.x. PMID 12786607
- [Background] Lewis BS, Eisen GM, Friedman S. A pooled analysis to evaluate results of capsule endoscopy trials. Endoscopy. 2005 Oct;37(10):960-5. doi: 10.1055/s-2005-870353. PMID 16189768
- [Background] Mow WS, Lo SK, Targan SR, Dubinsky MC, Treyzon L, Abreu-Martin MT, Papadakis KA, Vasiliauskas EA. Initial experience with wireless capsule enteroscopy in the diagnosis and management of inflammatory bowel disease. Clin Gastroenterol Hepatol. 2004 Jan;2(1):31-40. doi: 10.1016/s1542-3565(03)00289-1. PMID 15017630
- [Background] Dray X, Vahedi K, Valleur P, Marteau P. Is there any need for video capsule endoscopy evaluation in postduodenal small-bowel polyps detection in familial adenomatous polyposis? Gastrointest Endosc. 2007 Sep;66(3):634; author reply 634-5. doi: 10.1016/j.gie.2007.04.008. No abstract available. PMID 17725961
- [Background] Dionisio PM, Gurudu SR, Leighton JA, Leontiadis GI, Fleischer DE, Hara AK, Heigh RI, Shiff AD, Sharma VK. Capsule endoscopy has a significantly higher diagnostic yield in patients with suspected and established small-bowel Crohn's disease: a meta-analysis. Am J Gastroenterol. 2010 Jun;105(6):1240-8; quiz 1249. doi: 10.1038/ajg.2009.713. Epub 2009 Dec 22. PMID 20029412
- [Background] van Assche G, Vermeire S, Rutgeerts P. Mucosal healing and anti TNFs in IBD. Curr Drug Targets. 2010 Feb;11(2):227-33. doi: 10.2174/138945010790309902. PMID 20210770
- [Background] D'haens G, Van Deventer S, Van Hogezand R, Chalmers D, Kothe C, Baert F, Braakman T, Schaible T, Geboes K, Rutgeerts P. Endoscopic and histological healing with infliximab anti-tumor necrosis factor antibodies in Crohn's disease: A European multicenter trial. Gastroenterology. 1999 May;116(5):1029-34. doi: 10.1016/s0016-5085(99)70005-3. PMID 10220494
- [Background] Hanauer SB, Feagan BG, Lichtenstein GR, Mayer LF, Schreiber S, Colombel JF, Rachmilewitz D, Wolf DC, Olson A, Bao W, Rutgeerts P; ACCENT I Study Group. Maintenance infliximab for Crohn's disease: the ACCENT I randomised trial. Lancet. 2002 May 4;359(9317):1541-9. doi: 10.1016/S0140-6736(02)08512-4. PMID 12047962
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Rutgeerts P, Diamond RH, Bala M, Olson A, Lichtenstein GR, Bao W, Patel K, Wolf DC, Safdi M, Colombel JF, Lashner B, Hanauer SB. Scheduled maintenance treatment with infliximab is superior to episodic treatment for the healing of mucosal ulceration associated with Crohn's disease. Gastrointest Endosc. 2006 Mar;63(3):433-42; quiz 464. doi: 10.1016/j.gie.2005.08.011. PMID 16500392
- [Background] Dubcenco E, Jeejeebhoy KN, Petroniene R, Tang SJ, Zalev AH, Gardiner GW, Baker JP. Capsule endoscopy findings in patients with established and suspected small-bowel Crohn's disease: correlation with radiologic, endoscopic, and histologic findings. Gastrointest Endosc. 2005 Oct;62(4):538-44. doi: 10.1016/j.gie.2005.06.026. PMID 16185968
- [Background] Postgate AJ, Burling D, Gupta A, Fitzpatrick A, Fraser C. Safety, reliability and limitations of the given patency capsule in patients at risk of capsule retention: a 3-year technical review. Dig Dis Sci. 2008 Oct;53(10):2732-8. doi: 10.1007/s10620-008-0210-5. Epub 2008 Mar 5. PMID 18320313
- See also: sponsor link — http://www.getaid.org